CLINICAL TRIAL: NCT06709898
Title: Stroke in Working Age and Job Accommodation in Facilitating Transition Back to Work
Acronym: SWIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: Helsinki University Central Hospital (Other); Finnish Work Environment Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4011001
Record Dates: First submitted 2024-11-19; First posted 2024-11-29 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Ischemic; Cognitive Impairment; Fatigability Post Stroke; Mood Disturbances
Keywords: Stroke; Cognitive impairment; Return to work; Job accommodation; Work ability; Neuropsychology
MeSH Terms: conditions — Ischemic Stroke; Cognitive Dysfunction; Stroke

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive job accommodation (Experimental): * In intervention neuropsychological information will be individually processed and transferred systematically from the neurological unit to occupational health service (OHS) to help design the individually tailored work modifications.
  * Information of the job accommodation will be given to employers.
  * Cognitive job accommodation is carried out at the workplace in cooperation between the employer, employee and OHS.
  * Feedback of the cognitively challenging work traits will be given to participants after returning to work.
  Interventions: Other: Cognitive job accommodation
- Reference group (No Intervention): Employees return to work according to standard health care and workplace procedures.

INTERVENTIONS:
Other: Cognitive job accommodation — Job accommodation focused on the cognitive aspects at work
  Arms: Cognitive job accommodation

SUMMARY:
The aim of this randomized controlled trial (RCT) is to investigate whether cognitive job accommodation intervention enhances return to work, work ability and performance after ischemic stroke in working-age population. The main questions are:

* Does the cognitive job accommodation intervention affect absenteeism and presenteeism after stroke?
* Does the intervention affect work ability and perceived cognitive and emotional difficulties at work?
* Does the intervention decrease mental strain, fatigue and negative mood symptoms after return to work?
* Does the intervention affect life satisfaction among the stroke patients returning to work?

Researchers will compare the intervention group to a control group returning to work after stroke with current healthcare practices and work procedures.

Participants:

* At baseline, 6 and 12 month follow-up web-based questionnaires and cognitive tests are administered.
* At 3 month follow-up participants fill in Brain Work Questionnaire (BWQ) that measures cognitive demands and difficulties at work.

DETAILED DESCRIPTION:
Introduction: Strokes are one of the most significant conditions affecting cognition among working-age adults. Incidence of stroke increases in older age and due to the lengthening of working careers, more people are experiencing strokes while still employed. Additionally, the incidence of strokes among younger workers has increased over recent decades. In Finland, 2000 - 3000 work-aged persons suffer a stroke annually. The majority experiences cognitive or emotional symptoms post-stroke, and for about half of them, these symptoms become long-lasting or permanent. The cognitive demands of modern work have steadily increased, and the severity of cognitive symptoms has been shown to strongly predict the likelihood of returning to work after a stroke. While job accommodation has been shown to be an effective way to support return to work after many illnesses, there is limited research on its benefits following a stroke. Furthermore, there is lack of research on cognitive job accommodation, despite health professionals finding it particularly challenging.

Aims: To evaluate the effect of job accommodations after stroke on various work and health related outcomes. In addition, information about working-aged stroke patients returning to work and the practices of job accommodation is provided. In the future these results can potentially be applied also to other conditions affecting cognition.

Participants and methods: This study will recruit 18-68 year old stroke patients who are returning to work (n ≈ 100). Participants will be randomized into either a job accommodation intervention group or a control group. The study will assess the benefits of cognitive job accommodation in terms of absenteeism, presenteeism, work modifications, perceived work ability, health indicators and cognitive and emotional symptoms. Participants will be followed through web-based surveys and novel cognitive tests over a 12-month period. The study will adopt a multidisciplinary approach (ergonomics, occupational psychology, neuropsychology, and medicine) and will be based on the International Classification of Functioning, Disability, and Health (ICF) model. Cognitive job accommodation will utilize an established model, a design form, and an instructional video.

Collaborators and target organizations: The research will be conducted in collaboration with the Helsinki University Hospital Neurocenter and the Finnish Institute of Occupational Health. In addition to these organizations the study is funded by the Finnish Work Environment Fund. The target organizations include occupational health services and workplaces of stroke survivors.

Utilization of Results: The methods developed in this study can be used in future collaborations between workplaces, occupational health services, and specialized healthcare. The findings can also be applied to other conditions that cause cognitive difficulties and require job accommodation.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke occurred within 12 month
* At least mild cognitive, emotional and/or state alertness symptoms detected in neuropsychological assessment in subacute phase
* Employed when the stroke occurred and has workplace where to return
* Occupational health services (OHS) available
* Participant has agreed that clinical neuropsychologist and researcher can participate to OHS consultation regarding the job accommodation
* Adequate Finnish language ability to the questionnaires and cognitive tests

Exclusion Criteria:

* Work status - professional driver or some other safety critical occupation where even mild cognitive impairments restrict return to work
* Former neurological or psychiatric disorder or developmental disability affecting significantly cognition

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Absenteeism and presenteeism | 6 and 12 months
  Absenteeism and presenteeism are evaluated with World Health Organization's Health and Work Performance Questionnaire (HPQ) using both absolute and relative measures. Absolute absenteeism: hours in 4 week (higher value indicates worse outcome). Absolute presenteeism: single question measure of own job performance (score 0-10) analyzed according to the HPQ instructions (higher value indicates better outcome). Relative absenteeism: working hours in 4 week / expected working hours in 4 week. Relative presenteeism: evaluation of own job performance (score 0-10) / evaluation of most other workers job performance (score 0-10). This score is restricted to the range of 0.25 to 2.0 according to HPQ instructions. In both relative scores higher values indicate better outcome.
Work ability | 6 and 12 months
  Estimate of the current work ability measured with single question (score range 0-10, higher score indicate better outcome) from Work Ability Index. Estimate of future work ability measured with single question (categorical variable: yes, no, maybe) from Work Ability Index.

SECONDARY OUTCOMES:
Perceived success in returning to work | 6 and 12 months
  Subjectively evaluated success in returning to work. Single item question with 5 point Likert scale (5= very good; 1= very bad).
Cognitive demands of work and related difficulties | 3 and 12 months
  Frequency of different cognitive demands at work and related perceived difficulties measured with Brain Work Questionnaire. Frequency values are reported as averaged occurrence/week (lower values indicate better outcome), and related difficulties in ordinal response variable (0=no difficulties, 1=sometimes difficult, 2=often difficult). Higher value indicates worse outcome.
Cognitive symptoms at work | 6 and 12 months
  Cognitive symptoms at work measured with The Cognitive Function at Work Questionnaire total score (score range 0-58: higher value indicates worse outcome)
Stress | 6 and 12 months
  Estimates of perceived stress. General stress measured with single item stress question (score range 1-5, lower value indicates better outcome). Theme specific stress (at home, work and financial). Ordinal 4 point response scales. Questions from INTERSTROKE study.
Sick leave days | 6 and 12 months
  Number of days on sick leave after returning to work. Higher value indicates worse outcome.
Insomnia symptoms | 6 and 12 months
  Frequency of insomnia symptoms measured with single item question with ordinal 5 point scale (5=Every night or nearly every night; 1=never). Higher value indicates worse outcome.
Fatigue symptoms | 6 and 12 months
  Fatigue symptoms measured with Fatigue Assessment Scale (FAS). Total score range 10-50. Higher score indicates worse outcome.
Stroke related life satisfaction | 6 and 12 months
  Perceived life satisfaction based on the Young Stroke Questionnaire (total score 0-100; where higher score indicates better outcome)
Mental job strain | 6 and 12 months
  Perceived mental job strain. Single item question with ordinal 1-5 point response scale (1=not at all; 5 very much). Higher value indicates worse outcome.
Perceived cognitive and emotional difficulties in general | 6 and 12 months
  Perceived cognitive and emotional difficulties in general measured with Check List for Cognitive and Emotional Consequences. Likert scale questions 0-2. Higher values indicate worse outcome.
Modified Rankin scale | 12 months from the stroke
  The Modified Rankin Scale (mRS) measures degree of disability/dependence after a stroke. The mRS is a 6 point disability scale with possible scores ranging from 0 to 5. Higher score indicates worse outcome.
Benefit of the job accommodations | 6 and 12 months
  Perceived benefit of the carried out job accommodations. Single item question with 5 point Likert scale (5=very much; 1=very little). Higher value indicates better outcome.
Job burnout symptoms | 6 and 12 months
  Job burnout symptoms measured with Burnout Assessment Tool (BAT) 4-item version. Averaged sum score: range 1-5. Higher score indicates worse outcome.
Depression symptoms | 6 and 12 months
  Depression symptoms measured with Patient health Questionnaire 9 question version (PHQ-9). Total score range 0-27. Higher score indicates worse outcome.
General life satisfaction | 6 and 12 months
  Perceived general life satisfaction measured with single item question with 5 point Likert scale (5=very satisfied; 1=very dissatisfied). Higher score indicates better outcome.
Daily function ability | 6 and 12 months
  Perceived daily ability to function measured with single item question (score range 0-10). Higher score indicates better outcome.
Amount of job accommodations | 6 and 12 months
  Amount of the actualized job accommodations measured with single item question. Ordinal 4 item scale. (3=A lot , 2=somewhat, 1=a little, 0=not at all). Higher value indicates better outcome.
Work participation | 6 and 12 months
  Monthly work participation percentage (%) as compared to fulltime working. Higher value indicate better outcome.

OTHER OUTCOMES:
Cognitive test performance | 6 and 12 months
  Performance in web-based cognitive tests measuring reaction time, attention, executive functions and verbal memory functions. Applied cognitive tests are Task Switching test and Verbal memory test (modified version of the RAVLT).
Level of social support | 6 and 12 months
  Self-reported level of social support measured with Oslo Social Support Scale 3-item version (OSSS-3). Sum score range 3-14. Higher score represent better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Teemu I Paajanen, Dr, Principal Investigator — Finnish Institute of Occupational Health
Locations (1):
- Helsinki University Hospital Stroke Unit, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
IPD not shared